CLINICAL TRIAL: NCT04610346
Title: Assessing an Animal-Assisted Treatment Program for Adults With Aphasia: The Persons With Aphasia Training Dogs Program
Acronym: PATD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sharon Antonucci, PhD, Director, MossRehab Aphasia Center, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2020-450; R03HD101146 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-30 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Aphasia
Keywords: aphasia; animal-assisted therapy
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two study arms, immediate or delayed treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Other): Participants in this group will begin the training protocol immediately (within 1 week) after baseline pre-training evaluation is completed.
  Interventions: Behavioral: Persons with Aphasia Training Dogs Program
- Delayed (Other): Participants in the delayed arm will participate in two pre-training evaluations, one immediately upon enrollment and one at the end of the delay period immediately before beginning training
  Interventions: Behavioral: Persons with Aphasia Training Dogs Program

INTERVENTIONS:
Behavioral: Persons with Aphasia Training Dogs Program — Participants will learn and apply positive reinforcement training techniques for working with dogs to train them in basic obedience behaviors (e.g., SIT, STAY).
  Other Names: PATD Program

SUMMARY:
The lives of more than 2 million Americans are affected by aphasia, an acquired language impairment most commonly resulting from stroke that affects the ability to remember and express words. The well-being of these individuals is affected not just by the loss of words that is aphasia, but also the loss of friendships and opportunities for community engagement in which the loss of words can result. This study evaluates an animal-assisted treatment, The Persons with Aphasia Training Dogs (PATD) Program, designed to target the psychosocial consequences of aphasia by training participants in positive reinforcement dog training techniques that harness new skill learning and the advantages of interaction with family- or shelter-dwelling dogs to increase confidence and social engagement to support participants in living well with aphasia.

DETAILED DESCRIPTION:
Our long-term goals are to evaluate the effectiveness of canine- assisted therapy for persons with aphasia (PWA) and to operationalize aphasia treatments targeting psychosocial consequences of aphasia such that they may be implemented with fidelity across clinical settings. The overall objective of this application is to determine the feasibility and impact of a canine-assisted therapy program, the Persons with Aphasia Training Dogs (PATD) Program. This feasibility study, a crucial first step toward our long-term goals, will evaluate participants' ability to learn positive reinforcement dog training techniques, and provide data regarding the impact of treatment with respect to feasibility metrics associated with recruitment, retention, compliance, and importantly, program satisfaction/acceptability. The hypotheses are that PWA are able to learn positive reinforcement techniques to apply to dog training and that retention, compliance, and program satisfaction rates for this canine-assisted treatment will be high, with program satisfaction linked to psychosocial benefits such as increased self-confidence and social engagement for PWA. These hypotheses have been formulated on the basis of the PI's funded work designing and implementing the PATD program for the MossRehab Aphasia Center, as well as work in aphasia rehabilitation and canine-assisted interventions, including those with persons with aphasia. Accomplishment of the overall objective of this application will be achieved through this small-scale feasibility study aimed to garner preliminary support for our hypotheses and provide data to inform design of a future, large-scale clinical trial.

Specific Aim 1: Determine whether PWA, through participation in the PATD program, can learn and implement positive reinforcement techniques to train dogs in basic obedience skills. Hypothesis 1: On program completion, PWA will be competent in using positive reinforcement techniques, to independently cue a dog to complete a minimum of 4 (of 5) trained obedience skills. To test this hypothesis, participants will be assessed using a PI-adapted version of the Pet Partners© Animal-Handler Evaluation.

Specific Aim 2: Define participant characteristics associated with recruitment, retention, compliance and program acceptability/satisfaction relevant for determining PATD candidacy. Hypothesis 2: PWA will demonstrate high (above 80%) retention and compliance rates, and high program satisfaction, including increases in self-reported ratings of psychosocial well-being. To test this hypothesis, our primary outcome measure will be the Assessment of Living with Aphasia, complemented by self-report of participants' PATD experience gathered through an ALA-modeled qualitative spoken interview and a written, aphasia-friendly, satisfaction survey.

Accomplishment of the overall objective of this application will be achieved through this small-scale, feasibility study aimed to garner preliminary support for our hypotheses and to provide the foundation for a future, large-scale clinical trial.

Specific Aim 1: Determine whether PWA, through participation in the PATD program, can learn and implement positive reinforcement techniques to train dogs in basic obedience skills. Hypothesis 1: On program completion, PWA will be competent in using positive reinforcement techniques, to independently cue a dog to complete a minimum of 4 (of 5) trained obedience skills. To test this hypothesis, program participants will be assessed using a PI-adapted version of the Pet Partners© Animal-Handler Evaluation.

Skills Training: In consultation with a certified professional dog trainer, the PATD program was developed by the PI, a trained speech language-pathologist with eighteen years of experience working with people with aphasia, who has spent more than ten years working with shelter animals using positive reinforcement techniques. Participants enrolled in the PATD program will engage in five once-weekly individual training sessions with the PI, either with a family dog (PATD) or by volunteering at a local shelter, the Pennsylvania SPCA (PATD-PSPCA). PATD-PSPCA participants will work only with dogs that have been evaluated by PSPCA staff as appropriate for interaction with new volunteers. Each session will be dedicated to one of five pre-determined, sequentially-presented, obedience skills (i.e., LOOK, TOUCH, SIT, STAY, COME). Training sessions will last approximately 75 minutes, with an additional half hour allotted to the beginning of the first training session to review principles of positive-reinforcement training. Subsequent sessions will begin with a brief probe of the participant's skill in cueing the dog to perform the behavior trained the previous week. Following the probe, sessions will continue with a review of that week's lesson plan, after which the PI will model the first training step three times. After the model has been provided, the participant will attempt the procedure, receiving instructive feedback or reinforcement from the trainer. Instruction will proceed to the subsequent step when the participant and dog have attained 5 successful trials at the current step. The same demonstration procedure will be used at each subsequent step. Commands will be trained using one hand gesture for each behavior. To mark behaviors, participants will use a clicker attached to a wrist band, which can be hand-held or allowed to dangle for ease of use for those with hemiplegia. Participants will have the option of introducing the verbal command, but will not be required to do so. All participants will be asked to provide their dog with a walk before training sessions to support the dog in being ready to participate.

Skills Practice: Participants will not be required to complete all steps for an obedience skill in a single session, and will be encouraged to practice the skill with the dog for at least 3 practice sessions over the course of the week. Practice will be used as a measure of participant compliance. Each participant will be provided with a copy of the lesson plan and, if interested, a video demonstrating the PI performing the target skill with her own dog. Participants will also be provided with a training log to complete after each time they practice over the course of the week. Using a nine-point visual analog scale adapted from the Assessment of Living with Aphasia (ALA), participants will rate their own and the dog's performance during each practice session. To facilitate responses on the log, participants will be provided with a pictographic list of questions to consider in determining their ratings (e.g., "How many times did I have to cue the dog", "Did I 'click' as soon as the dog did what I asked?".

Specific Aim 2: Define participant characteristics associated with recruitment, retention, compliance and program acceptability/satisfaction relevant for determining PATD candidacy. Hypothesis 2: PWA will demonstrate high (above 80%) retention and compliance rates, and high program satisfaction, including increases in self-reported ratings of psychosocial well-being. To test this hypothesis, the primary outcome measure will be the Assessment of Living with Aphasia, complemented by self-report of participants' PATD experience gathered through an ALA-modeled qualitative spoken interview and a written, aphasia-friendly, satisfaction survey.

Feasibility Metrics: Recruitment rates will be tracked appropriate to the creation of a CONSORT flow diagram including: # contacted, # screened, # eligible (vs. ineligible), # consented/enrolled (vs. declined). To evaluate further the size of the population that may benefit from the treatment, participant screening will include surveying of interest in interaction with dogs and in dog-related activities. Similarly, participant retention rates will be tracked including: # completing baseline assessment, # completing immediate post-treatment assessment, and # completing follow-up assessment. Participant withdrawals will be tracked for whether initiated by researcher or participant. Participant compliance rates will be tracked including # assessment and training sessions (relative to total possible) completed, and # self-reported home practice sessions.

Outcome Measurement: The primary quantitative outcome measure of acceptability, the ALA, is a pictographic self-report measure of quality of life developed to assess the impact of aphasia on daily life. Questions address participants' perceptions of aphasia, their environment, their relationships, their community engagement, experiences of self-confidence and respect, and their progress toward "living well with aphasia". Participants respond by pointing to a visual analog scale, providing for quantification of responses, and rendering the tool accessible to those with language impairment. Overall score and subdomain scores have demonstrated acceptable-to-high test-retest reliability and internal consistency. To augment standardized evaluation, the PI has developed a complementary interview, consistent with the format of the ALA, to more specifically probe PATD participants' perceptions of the impact of the training program. Participant narratives produced during the administration will be supported using interviewing strategies appropriate for persons with aphasia. A written, visual analog scale satisfaction survey designed to adhere to guidelines of 'aphasia-friendly' written materials will also be administered. It is anticipated that the assessment battery will take two hours to complete.

Outcome Measurement/Participation Timeline: Participants will be randomized into immediate and waitlist treatment groups using permuted block randomization with stratification. Analysis between these two arms will be exploratory only in nature, and will inform us regarding the feasibility of the waitlist control design for use in a larger clinical trial. All participants will be evaluated before training begins, immediately following training, and at a 3-month follow-up. Participants in the delayed arm will participate in two pre-training evaluations, one immediately upon enrollment and one at the end of the delay period immediately before beginning training.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of aphasia acquired as the result of cerebro-vascular accident (CVA)
2. English as a native or primary language
3. Evidence of linguistic and cognitive capacity to understand the research requirements
4. Willingness and stamina to participate in the protocol
5. Lives within 1 hour driving distance to MRRI (50 Township Line Rd, Elkins Park, PA 19027 and (as appropriate) PSPCA HQ (350 E. Erie Ave., Philadelphia, PA 19134

Exclusion Criteria:

• Diagnosis of neurological injury or disease other than CVA

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Antonucci, Ph.D., Principal Investigator — AEHN
Locations (1):
- Moss Rehabilitation Research Institute, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams, D. L. (1997). Animal-assisted enhancement of speech therapy: A case study. Anthrozoös: A multidisciplinary journal of the interactions of people and animals, 10(1), 53-56.
- [Background] Beetz, A. M. (2017). Theories and possible processes of action in animal-assisted interventions. Applied Developmental Science, 21(2), 139-149.
- [Background] Hediger K, Thommen S, Wagner C, Gaab J, Hund-Georgiadis M. Effects of animal-assisted therapy on social behaviour in patients with acquired brain injury: a randomised controlled trial. Sci Rep. 2019 Apr 9;9(1):5831. doi: 10.1038/s41598-019-42280-0. PMID 30967589
- [Background] Hilari K, Needle JJ, Harrison KL. What are the important factors in health-related quality of life for people with aphasia? A systematic review. Arch Phys Med Rehabil. 2012 Jan;93(1 Suppl):S86-95. doi: 10.1016/j.apmr.2011.05.028. Epub 2011 Nov 25. PMID 22119074
- [Background] LaFrance C, Garcia LJ, Labreche J. The effect of a therapy dog on the communication skills of an adult with aphasia. J Commun Disord. 2007 May-Jun;40(3):215-24. doi: 10.1016/j.jcomdis.2006.06.010. Epub 2006 Sep 6. PMID 16950329
- [Background] Macauley BL. Animal-assisted therapy for persons with aphasia: A pilot study. J Rehabil Res Dev. 2006 May-Jun;43(3):357-66. doi: 10.1682/jrrd.2005.01.0027. PMID 17041821
- [Background] Shadden, B. (2005). Aphasia as identity theft: Theory and practice. Aphasiology, 19(3-5), 211-223

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants consented to participation either with a family dog or at a local animal shelter. People in the shelter dog condition were required to complete volunteer onboarding before beginning study activities. Five people consented to the shelter-dog condition were not able to complete shelter volunteer onboarding. They were withdrawn from the study prior to initiating study activities as they did not have access to a dog.
Period: Overall Study
Arm/Group | Immediate | Delayed
Started (Participants consented to participation either with a family dog or at a local animal shelter. People in the shelter dog condition were required to complete volunteer onboarding before beginning study activities. Five people consented to the shelter-dog condition were not able to complete shelter volunteer onboarding. They were withdrawn from the study prior to initiating study activities as they did not have access to a dog.) | 12 | 5
Mid-point (Evaluation Immediately After Training) | 9 | 3
Completed | 9 | 3
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — did not complete shelter onboarding | 2 | 1

BASELINE CHARACTERISTICS:
Population: Participants consented to participation either with a family dog or at a local animal shelter. People in the shelter dog condition were required to complete volunteer onboarding before beginning study activities. Five people consented to the shelter-dog condition were not able to complete shelter volunteer onboarding. They were withdrawn from the study prior to initiating study activities.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate | Delayed | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.67 (8.96) | 53.33 (12.1) | 60.33 (10.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 9 | 3 | 12
Western Aphasia Battery- Revised (WAB-R) [Mean (Standard Deviation); unit: units on a scale] — A standardized aphasia battery that provides a description of aphasia type and severity indicated by aphasia quotient (AQ), a criterion measures on a scale of 0-100 (0= most severe). Ranges of severity classified by the AQ are: 0-25 very severe aphasia; 26-50 severe aphasia; 51-75 moderate aphasia; and ≥76, mild aphasia to 'non-aphasic' per WAB.
  units on a scale | 89.6 (10.5) | 64.5 (35.9) | 83.3 (21.1)
Assessment of Living with Aphasia (ALA) [Mean (Standard Deviation); unit: units on a scale] — The ALA is a pictographic self-reported measure of quality of life living with aphasia across 4 domains (aphasia, participation, environment, and personal) as well as responding to how well they feel they are overcoming the 'wall' (obstacle) of aphasia. Participants respond using a visual-analog scale (0-4, 0= negative valence).
  For those in the delayed condition, the 2nd baseline (closest in time to treatment initiation) is reported. The delayed condition was primarily used to assess feasibility of the design for a future larger-scale clinical trial.
  units on a scale | 2.2 (0.6) | 2.2 (0.057) | 2.2 (0.5)
Confidence after Stroke Measure (CaSM) [Mean (Standard Deviation); unit: units on a scale] — The CaSM is a self-report measure that assesses three aspects of confidence after stroke, self-confidence, positive attitude, and social confidence. Participants self-rate on scales, with total values 0-81. Higher scores are associated with higher levels of confidence.
  For those in the delayed condition, the 2nd baseline (closest in time to treatment initiation) is reported. The delayed condition was primarily used to assess feasibility of the design for a future larger-scale clinical trial.
  units on a scale | 46.9 (7.9) | 52 (5.57) | 48.17 (7.52)
Behavioural Assessment of Dysexecutive Syndrome (BADS) [Mean (Standard Deviation); unit: units on a scale] — The BADS is a standardized assessment of executive function. Total profile scores range between 0-24, with higher scores being associated with more accurate performance. This measure was used for exploratory purposes. It has not been validated for use with individuals with aphasia and performance may be confounded by language difficulties associated with aphasia.
  For those in the delayed condition, the 2nd baseline (closest in time to treatment initiation) is reported. The delayed condition was primarily used to assess feasibility of the design for a future larger-scale clinical trial.
  units on a scale | 13.7 (4.2) | 13 (4.6) | 13.5 (4.1)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Living With Aphasia (ALA, Kagan et al., 2010)
Description: The Assessment of Living with Aphasia is a pictographic self-reported measure of quality of life living with aphasia across four domains (aphasia, participation, environment, and personal) and an overall evaluation of how well the participant judges that they are overcoming the 'wall' (obstacle) of aphasia. Participants respond using a visual-analog scale with nine points (0 (minimum), .5, 1, 1.5, 2, 2.5, 3, 3.5, 4 (maximum) with higher values being associated with a better outcome. The total scaled score (0- minimum - 4- maximum) is the sum of the raw scores in each of the four domains divided by the number of questions pertaining to each domain, plus the response to the 'wall' question.
Time Frame: Once within approximately 1 week of the end of training, then once approximately 3 months after end of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 9 | 3
units on a scale
  Immediately after Training | 2.67 (0.67) | 2.33 (0.06)
  Three months after training | 2.68 (0.69) | 2.43 (0.23)

2. Primary Outcome: PI-adapted Version of Pet Partners Animal-handler Evaluation.
Description: Participants were score on a PI-adapted version of the Pet Partners Animal-Handler Evaluation. Each participant was scored on a 3-point scale ( 0= not ready (minimum), 1= ok, 2= best (maximum)) by a certified professional dog trainer on their cueing of each of five basic obedience behaviors (LOOK, TOUCH TARGET, SIT, STAY, COME), hence the maximum score on each summative evaluation is 10 (rating of 2 x each of the 5 obedience behaviors). On this scale, a higher number indicates a better outcome. An a-priori criterion was set at 5 (out of 10) or higher for achieving competence.
Time Frame: Once within approximately 1 week of the end of training, then once approximately 3 months after end of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 9 | 3
units on a scale
  Immediately after training | 8.8 (1.2) | 5.3 (5.0)
  Three months after training | 9.2 (1.1) | 8 (3.5)

3. Secondary Outcome: The Confidence After Stroke Measure (Horne et al., 2017)
Description: The Confidence after Stroke Measures is a self-report measure that assesses three aspects of confidence after stroke, self-confidence, positive attitude, and social confidence. Per Horne et al., (2017) Participants self-rate on scales, with total values 0-81:
  Scale One -Self - Confidence = 0-27 Scale Two -Positive Attitude =0-24 Scale Three -Social Confidence =0-30
  Higher scores are associated with higher levels of confidence. A change on total score of 4 or more is reported as being considered clinically significant. A score of 36 (-1 SD) indicates a possible concern, a score of 28(-2 SD) indicates a probable problem.
Time Frame: Once within approximately 1 week of the end of training, then once approximately 3 months after end of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 9 | 3
units on a scale
  Immediately after training | 47.7 (9.7) | 55.67 (7.6)
  Three months after training | 49.4 (13.9) | 51.3 (7.4)

4. Secondary Outcome: Behavioural Assessment of Dysexecutive Syndrome (BADS) (Wilson et al., 1996)
Description: The Behavioral Assessment of Dysexecutive Syndrome is a standardized assessment of executive function that evaluates skills including planning, organization, and problem-solving. Total profile scores range between 0 (min) - 24 (max), higher scores are associated with a better outcome, i.e., more accurate performance. Total profile scores comprise sub-scores from six subtests:
  Temporal judgement - ability to estimate how long to complete various activities of daily life events.
  Rule shift cards - ability to change an established pattern of responding Action program - practical problem solving. Key search - strategy formation. Zoo map - planning. Modified six elements - planning, task scheduling and performance monitoring. Complete details are available in the BADS manual. This measure was used for exploratory purposes. It has not been validated for use with individuals with aphasia and performance may be confounded by language difficulties associated with aphasia.
Time Frame: Once within approximately 1 week of the end of training, then once approximately 3 months after end of training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate | Delayed
Number analyzed (Participants) | 9 | 3
units on a scale
  Immediately after training | 14.22 (5.56) | 16.7 (3.5)
  Three months after training | 15.3 (4.0) | 17.3 (3.8)

ADVERSE EVENTS:
Time Frame: Participants were monitored from baseline evaluation through followup evaluation. For individuals in the immediate condition this comprised approximately 19 weeks, whereas for those in the delayed condition this comprised approximately 25 weeks.
Description: Adverse events were defined consistent with clinicaltrials.gov definitions.
Arm/Group | Immediate | Delayed
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 0/9 | 0/3

LIMITATIONS AND CAVEATS:
Challenges to feasibility, both with respect to initial recruitment and completion (for those in the shelter dog condition) primarily related to access to a dog, not inability to engage in the treatment. However, we do not feel this unduly limits the feasibility of the treatment overall as future iterations are planned to be embedded within direct clinical service delivery with therapy or facility dog- handler teams, rather than relying on participants' own family dogs or shelter dogs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (5):
  • Study Protocol and Statistical Analysis Plan (2024-10-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT04610346/Prot_SAP_000.pdf
  • Informed Consent Form: Family Dog Immediate (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04610346/ICF_001.pdf
  • Informed Consent Form: Shelter Dog Immediate (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04610346/ICF_002.pdf
  • Informed Consent Form: Family Dog Delayed (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04610346/ICF_003.pdf
  • Informed Consent Form: Shelter Dog Delayed (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT04610346/ICF_004.pdf